CLINICAL TRIAL: NCT01475188
Title: Regulatory Lymphocytes (Treg) in the Modulation of Allergic Inflammation in Patients Treated With Specific Immunotherapy.
Brief Title: Regulatory Lymphocytes in Patients Treated With Specific Immunotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Pawel Gorski, prof, MD, PhD, Ministry of Science and Higher Education, Poland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: N 402 057 32/1788; 1788/PO1/2007/32 (Other Grant/Funding Number: Ministry of Science and Higher Education)
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Immunotherapy; Seasonal Allergic Rhinitis
Keywords: specific subcutaneous immunotherapy; seasonal allergic rhinitis; regulatory lymphocytes; signal transduction; histamine receptor
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — allergovit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): 20 patients with intermittent allergic rhinitis sensitized to grass pollen allergens
  Interventions: Other: placebo
- Specific subcutaneous immunotherapy (Active Comparator): 21 symptomatic patients with intermittent allergic rhinitis sensitized to grass pollen allergens
  Interventions: Drug: Allergovit

INTERVENTIONS:
Drug: Allergovit — commercially available grass pollen allergoid (100%), concentration A (1000 TU/ml, therapeutic units/ml)concentration B (10000 TU/ml).Patients were given subcutaneous injections with initial dose of 0.1 ml (concentration A) was increased once a 7 (+7) days until the highest tolerated dose (0.6, concentration B) was reached and SIT was continued with injections once every 4 - 6 weeks up to two years.
  Other Names: Allergovit, grass pollen 100%, Allergopharma, Germany
  Arms: Specific subcutaneous immunotherapy
Other: placebo — placebo administered with the same scheme and doses as specific subcutaneous immunotherapy
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether specific subcutaneous immunotherapy affects fractions of regulatory T lymphocytes and histamine H2 receptor expression and ZAP70 in regulatory T lymphocytes.

DETAILED DESCRIPTION:
Allergy constitutes an important problem worldwide thus effective treatment is crucial for the reduction of symptoms severity, patients' activity and quality of life as well as for the reduction of direct and indirect costs of the disease. Specific allergen immunotherapy (SIT) is a potentially curative and specific method of treatment for allergic diseases, particularly for intermittent allergic rhinitis. Specific subcutaneous immunotherapy induce peripheral tolerance and suppress inflammation in tissue. In periphery, effector T cells unresponsiveness to antigens is mediated mainly by allergen specific regulatory T cells. Regulatory T cells induced peripherally comprise IL-10 producing type 1 regulatory T cells (Tr1) and regulatory T cells subset arising in vitro from CD4+CD25- and in vivo from peripheral memory T cells whereas naturally occurring Tregs (nTregs)originate in thymus and represent about 5% of the peripheral CD4 T cells and constitutively express high levels of the high-affinity IL-2 receptor (CD25hi). They coexpress Forkhead Box Protein P3 (Foxp3), glucocorticoid induced tumor necrosis factor receptor (GITR), cytotoxic T lymphocyte associated antigen (CTLA-4), and display low expression of alpha chain of the IL-7 receptor. Although clinical and immunological outcomes of SIT, that are associated with regulatory T cells functions were profoundly studied, little is known about the molecular mechanisms that are crucial for nTregs activation and function in the course of SIT. Since histamine is a key mediator in allergy that exerts its effect through 4 types of histamine receptors we decided to investigate the expression of histamine 2 receptor, that has potent immunomodulatory properties, in regulatory lymphocytes in patients treated with SIT. Furthermore, since T cell receptor activation is essential for T effector lymphocytes activation we wanted to check the expression of zeta chain associated protein (ZAP70), that constitutes a linker between TCR and lower levels of intracellular downstream signal transduction, in regulatory T cells in the course of SIT.

This is a 3-year prospective, placebo controlled, double blind trial of grass SIT. 41 patients with seasonal allergic rhinitis were randomized to receive SIT (n = 21) or placebo (n = 20) and 15 healthy were included as a control. The primary and secondary outcomes were assessed at baseline and during the treatment period - before the start of the pollen season, at the height of the pollen season and after the end of the pollen season.Results were compared between the treatment year and baseline and between the groups treated with SIT, placebo and healthy control.

ELIGIBILITY:
Inclusion Criteria:

* seasonal allergic rhinitis with or without allergic conjunctivitis
* sensitization to grass pollen allergens (confirmed with skin prick tests, conjunctival provocation test, specific IgE)
* symptoms of allergic rhinitis with or without conjunctivitis for at least 2 years before the study

Exclusion Criteria:

* sensitization to allergens, that could interfere with grass pollen
* asthma
* cystic fibrosis
* ciliary dysmotility syndrome
* bronchiectasis
* smoking
* tuberculosis
* neoplastic disease
* chronic sinusitis and nasal polyps
* systemic glucocorticosteroids treatment
* treatment with immunotherapy in the past

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
numbers of regulatory T lymphocytes (nTregs) | Change from the baseline year to the 2nd year of immunotherapy.
  Numbers of regulatory T cells (nTregs) at baseline year both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen season and in the 2nd year of immunotherapy both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen.

SECONDARY OUTCOMES:
Expression of zeta chain associated protein (ZAp70) in regulatory lymphocytes (nTregs) | Change from the baseline year to the 2nd year of immunotherapy
  Expression of zeta chain associated protein (ZAP70) in regulatory T cells (nTregs) at baseline year both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen season and in the 2nd year of immunotherapy both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen.
Expression of histamine H2 receptor in regulatory lymphocytes (NTregs) | Change from the baseline year to the second year of immunotherapy
  Expression of histamine H2 receptor in regulatory T cells (nTregs) at baseline year both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen season and in the 2nd year of immunotherapy both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen.
Rhinoconjunctivitis symptom score | Change from the baseline year to the second year of immunotherapy
  Change of the rhinoconjunctivitis symptoms score from the baseline year to the 2nd year of immunotherapy
Nasal eosinophilia | Change from the basline year to the 2nd year of immunotherapy
  Numbers of eosinophils in nasal lavage during the baseline year both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen season and in the 2nd year of immunotherapy both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen.
Concentration of nitric oxide in exhaled air | Change from the baseline year to the 2nd year of immunotherapy
  Concentration of nitric oxide in exhaled air during the baseline year both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen season and in the 2nd year of immunotherapy both 6 weeks before the start of the pollen season, at the height of pollen season and 6 weeks after the termination of the pollen.
Consumption of rescue medications | Change from the baseline year to the second year of imunotherapy
  Comparison of the rescue medication intake during the baseline year and during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Górski, Prof, MD, PhD, Study Chair — Department of Pneumonology and Allergy, Medical University of Lodz, Poland
Locations (1):
- Department of Pneumonology and Allergy, Medical University of Lodz, Lodz, Poland

REFERENCES:
- [Background] Dieckmann D, Bruett CH, Ploettner H, Lutz MB, Schuler G. Human CD4(+)CD25(+) regulatory, contact-dependent T cells induce interleukin 10-producing, contact-independent type 1-like regulatory T cells [corrected]. J Exp Med. 2002 Jul 15;196(2):247-53. doi: 10.1084/jem.20020642. PMID 12119349
- [Background] Baecher-Allan C, Viglietta V, Hafler DA. Human CD4+CD25+ regulatory T cells. Semin Immunol. 2004 Apr;16(2):89-98. doi: 10.1016/j.smim.2003.12.005. PMID 15036232
- [Background] Fontenot JD, Gavin MA, Rudensky AY. Foxp3 programs the development and function of CD4+CD25+ regulatory T cells. Nat Immunol. 2003 Apr;4(4):330-6. doi: 10.1038/ni904. Epub 2003 Mar 3. PMID 12612578
- [Background] Cao D, Malmstrom V, Baecher-Allan C, Hafler D, Klareskog L, Trollmo C. Isolation and functional characterization of regulatory CD25brightCD4+ T cells from the target organ of patients with rheumatoid arthritis. Eur J Immunol. 2003 Jan;33(1):215-23. doi: 10.1002/immu.200390024. PMID 12594850
- [Background] Sakaguchi S. Naturally arising CD4+ regulatory t cells for immunologic self-tolerance and negative control of immune responses. Annu Rev Immunol. 2004;22:531-62. doi: 10.1146/annurev.immunol.21.120601.141122. PMID 15032588
- [Background] Jordan MS, Riley MP, von Boehmer H, Caton AJ. Anergy and suppression regulate CD4(+) T cell responses to a self peptide. Eur J Immunol. 2000 Jan;30(1):136-44. doi: 10.1002/1521-4141(200001)30:13.0.CO;2-0. PMID 10602035
- [Background] Apostolou I, Sarukhan A, Klein L, von Boehmer H. Origin of regulatory T cells with known specificity for antigen. Nat Immunol. 2002 Aug;3(8):756-63. doi: 10.1038/ni816. Epub 2002 Jul 1. PMID 12089509
- [Background] Hori S, Nomura T, Sakaguchi S. Control of regulatory T cell development by the transcription factor Foxp3. Science. 2003 Feb 14;299(5609):1057-61. doi: 10.1126/science.1079490. Epub 2003 Jan 9. PMID 12522256
- [Background] Shevach EM. CD4+ CD25+ suppressor T cells: more questions than answers. Nat Rev Immunol. 2002 Jun;2(6):389-400. doi: 10.1038/nri821. PMID 12093005
- [Background] Thornton AM, Shevach EM. CD4+CD25+ immunoregulatory T cells suppress polyclonal T cell activation in vitro by inhibiting interleukin 2 production. J Exp Med. 1998 Jul 20;188(2):287-96. doi: 10.1084/jem.188.2.287. PMID 9670041
- [Background] Fontenot JD, Rasmussen JP, Williams LM, Dooley JL, Farr AG, Rudensky AY. Regulatory T cell lineage specification by the forkhead transcription factor foxp3. Immunity. 2005 Mar;22(3):329-41. doi: 10.1016/j.immuni.2005.01.016. PMID 15780990
- [Background] Jutel M, Akdis M, Blaser K, Akdis CA. Mechanisms of allergen specific immunotherapy--T-cell tolerance and more. Allergy. 2006 Jul;61(7):796-807. doi: 10.1111/j.1398-9995.2006.01175.x. PMID 16792576
- [Background] Jutel M, Watanabe T, Klunker S, Akdis M, Thomet OA, Malolepszy J, Zak-Nejmark T, Koga R, Kobayashi T, Blaser K, Akdis CA. Histamine regulates T-cell and antibody responses by differential expression of H1 and H2 receptors. Nature. 2001 Sep 27;413(6854):420-5. doi: 10.1038/35096564. PMID 11574888
- [Background] Liu H, Rhodes M, Wiest DL, Vignali DA. On the dynamics of TCR:CD3 complex cell surface expression and downmodulation. Immunity. 2000 Nov;13(5):665-75. doi: 10.1016/s1074-7613(00)00066-2. PMID 11114379
- [Derived] Ciebiada M, Kasztalska K, Gorska-Ciebiada M, Gorski P. ZAP70 expression in regulatory T cells in allergic rhinitis: effect of immunotherapy. Clin Exp Allergy. 2013 Jul;43(7):752-61. doi: 10.1111/cea.12124. PMID 23786282